CLINICAL TRIAL: NCT06382194
Title: Shared Decision Making for Firearm Safety Among Older Adults With Early Changes Associated With Alzheimer's Disease/Alzheimer's Disease-Related Dementias (AD/ADRD)
Brief Title: Decision Making Tool for Firearm Storage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Phelan, Professor, Division of Gerontology and Geriatric Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00014522; 1R21AG076362-01 (NIH)
Record Dates: First submitted 2024-04-02; First posted 2024-04-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Dementia, Mild; Depression
MeSH Terms: conditions — Dementia; Lymphoma, Follicular; Depression | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Participants in this arm will receive the intervention and undergo research assessments.
  Interventions: Other: Decision aid

INTERVENTIONS:
Other: Decision aid — The intervention is a newly developed decision aid designed to guide decisions about storage of firearms among older gun owners with early dementia and/or depression.

SUMMARY:
This is a one-arm pilot study testing the feasibility and acceptability of a decision aid about safe firearm storage.

DETAILED DESCRIPTION:
This pilot study will test the feasibility and acceptability of a decision aid about safe firearm storage with firearm-owning persons with early dementia and/or depression

ELIGIBILITY:
Inclusion Criteria:

* Medical record documentation of early dementia and/or depression
* Internet or mobile device access
* Access to firearm(s)

Exclusion Criteria:

• Active suicidality

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Firearm storage (adapted from the National Firearm Survey) | Assessed at 4 weeks post enrollment
  An ordinal measure of how firearms are stored (from relinquishment to loaded/unlocked)

SECONDARY OUTCOMES:
Low-Literacy Decisional Conflict Scale | Assessed at 4 weeks post enrollment
  Measured by the Low Literacy Decisional Conflict Scale. This is a 10-item scale comprised of 4 subscales. Response options for each item are yes, no, unsure. Score range is from 0 (no decisional conflict) to 100 (extremely high decisional conflict).
Knowledge Questionnaire | Assessed at 4 weeks post enrollment
  A measure of participant understanding of firearm safe storage, alternatives, rationale, risks and benefits. Each item is given a score value of 1 (if participant correctly selects 'true' or 'false') or zero (if selects the incorrect answer or selects 'unsure'). Items are totaled to obtain an overall knowledge score.
Feasibility of intervention delivery | Assessed at 4 weeks post enrollment
  Number of participants who access and view the entire decision aid
Acceptability of Intervention Measure | Assessed at 4 weeks post enrollment
  A 4-item measure of the intervention's acceptability. The response option for each item is a 5-point Likert scale, ranging from 1 (completely disagree) to 5 (completely agree).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Phelan, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States